CLINICAL TRIAL: NCT06950203
Title: A Randomised, Double Blinded Study to Determine the Effect of Supplementation With Fish Oil (EPAX EVOLVE 05) on Sperm Quality in Healthy Men.
Brief Title: The Effect of Supplementation With Fish Oil (EPAX EVOLVE 05) on Sperm Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Epax Norway AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: VLC 2024 01 Fertility
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Infertility, Male
Keywords: VLCFA; VLC-PUFA; Very long chain polyunsaturated fatty acids; fertility; supplement
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Active Comparator): DHA fish oil to match DHA content in active arm
  Interventions: Dietary Supplement: Comparator arm (DHA)
- VLC-PUFA (Experimental): EPAX EVOLVE 05 containing Very Long Chain Polyunsaturated Fatty Acids
  Interventions: Dietary Supplement: Very Long Chain Polyunsaturated Fatty Acids

INTERVENTIONS:
Dietary Supplement: Very Long Chain Polyunsaturated Fatty Acids — Fish oil with DHA and VLCPUFA
  Arms: VLC-PUFA
Dietary Supplement: Comparator arm (DHA) — Oil containing equal DHA content to active arm
  Arms: Placebo

SUMMARY:
The study will enrol men that have a poor sperm quality. They will take either a placebo or fish oil capsule (2 per day) for 3 months. At the beginning and end of the study the participant will be asked for a sperm sample for measuring quality parameters.

DETAILED DESCRIPTION:
The study is a 2-armed, comparator controlled, double-blinded study. Subjects, study staff, sperm quality assessor and statistician will be blinded to the nutritional intervention.

The study Sponsor will be unblinded for purposes of packaging and supply of nutritional products.

Screening (Visit 0). Subjects will be asked to join the study based on an analysis documenting poor semen quality. Subjects will be informed about the result of the semen analysis and informed that the clinic is participating in a study about sperm quality. Subjects that show interest to participate will be verbally and in writing given further information about the study and the study procedures by dedicated study personnel. Patients willing to sign the consent will have the possibility to ask further questions. The clinic will provide a screening log with restricted access, containing screening number and subject identification.

Enrolment (Visit 1). For eligible subjects, the study coordinator will take the consent on behalf of the clinic.

Subjects who satisfy all inclusion criteria and no exclusion criteria will be randomised to investigational product or comparator and given a randomisation number and will receive enough capsules for 12 weeks. The clinic will provide a randomization log with non-identifiable information.

Telephone follow-up (Visit 2). After 6 weeks (± 1 week), a dedicated study nurse will contact the subject by phone. During the call, subjects will be asked about their well-being, whether they have been consistently taking their capsules, and if they are experiencing any issues that may be related to the study product.

Final Visit (Visit 3). 12 weeks (± 1 week) after the study commencement, the subject will attend a follow-up physical visit and return any remaining capsules.

Subjects will be examined for vital signs, physical examination, relevant medical history, current medications, smoking and alcohol habits and a food frequency questionnaire. A period of abstinence (2 days) will be requested prior to study specific sperm samples.

Each subject will take 2 x 1.0g capsules of EVOLVE 05 daily for 3 months or 2 x 1.0g comparator capsules.

Sperm samples for quality measurements will be taken at visit 1 and visit 3. The remaining sample will be frozen and maintained for analysis of VLCFA content.

Dietary intake will be recorded to control for marine specific dietary variables: Assessment at visit 1 and visit 3 using a brief questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18-55
2. Referred for or claiming a semen analysis.
3. Willing to have at least 2 days abstinence of sexual activity prior to a sperm sample being taken.
4. Reduced semen quality defined as:

   • Progressive motility: <30%
5. Willing to refrain from omega-3/cod liver oil supplementation during the study. Use of other supplements is allowed.

   -

Exclusion Criteria:

1. Known allergy to fish products
2. Historically, known, or suspected bacterial infection in reproductive organs
3. Varicocele suspected from physical examination
4. Azoospermia
5. Diagnosis of diabetes (type 2)
6. Diagnosis of Crohn´s Disease
7. Inferior semen quality due to medical reasons, such as cryptorchidism (via questionnaire/medical records) -

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Males
Enrollment: 80 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Total Progressive Motile count will be measured pre- and post-intervention and compared to the comparator arm. | From baseline to end of intervention at 3 months
  The motile count will be performed by competent operators at each clinical site.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicus Group AS, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data may be shared on request from relevant academics.